CLINICAL TRIAL: NCT00073710
Title: A Phase IV, Single-Center, Active-Controlled Cross-Over Pilot Study to Evaluate the Effects of Zemplar Injection and Calcijex on Intestinal Absorption of Calcium
Brief Title: Study to Evaluate the Effects of Zemplar Injection and Calcijex on Intestinal Absorption of Calcium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M01-375
Record Dates: First submitted 2003-12-03; First posted 2003-12-04 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: secondary hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — paricalcitol; Calcitriol

INTERVENTIONS:
Drug: Zemplar
Procedure: 42 Ca carbonate absorption via single tracer method
Drug: Calcijex

SUMMARY:
A study to investigate the effects of Zemplar and Calcijex on intestinal calcium absorption in hemodialysis subjects.

ELIGIBILITY:
Inclusion Criteria

* Subject is ≥ 20 years of age.
* Subject is diagnosed with ESRD, and must be on maintenance hemodialysis (HD) three times a week for at least 2 months prior to the Screening Phase and expected to remain on HD for the duration of the study.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

  * Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
  * Contraceptives (oral or parenteral) for three months prior to study drug administration
  * In a monogamous relationship with a vasectomized partner
* If female, subject is not breastfeeding and has a negative serum pregnancy test prior to the treatment phase.
* Subject had an intact PTH value > 200 pg/mL.
* Serum calcium level < 10.2 mg/dL at Screening visit.
* Serum phosphorus level < 6.5 mg/dL at Screening visit.
* Ca´P product ≤ 65 at Screening visit.
* Must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the conduct of any study-specific procedure

Exclusion Criteria

* Subject has a history of an allergic reaction or significant sensitivity to vitamin D or vitamin D related compounds.
* Subject has chronic gastrointestinal disease, which in the Investigator's opinion, may result in clinically significant GI malabsorption.
* Liver function defects defined as > 2 times the upper limit of normal for liver enzyme or > 1.5 times the upper limit of normal coagulation levels.
* Subject is taking maintenance calcitonin, glucocorticoids in an equivalent dose > 5 mg prednisone, or other drugs that may affect calcium or bone metabolism, other than females on stable (same dose and product for 3 months) estrogen and/or progestin therapy.
* For any reason, subject is considered by the Investigator to be an unsuitable candidate to receive pharmacological doses of vitamin D.
* Subject has received any investigational drug within 4 weeks prior to the Treatment Phase.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-09

PRIMARY OUTCOMES:
The mean within subject difference in calcium absorption rates between treatment regimens will be analyzed using ANOVA appropriate for a two-period cross-over trial.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lund, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States